CLINICAL TRIAL: NCT07066670
Title: Comparative Effects of Strain Counterstrain and Muscle Energy Technique on Pain, Range of Motion, and Functional Disability in Patients of Knee Osteoarthritis
Brief Title: Strain Counterstrain and Muscle Energy Technique in Patients of Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Iqra zahid, Student, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rec-UOL-/204/08/24
Record Dates: First submitted 2025-04-03; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: Knee Osteoarthritis; Strain Counterstrain; Muscle Energy Technique; Pain Management; Functional Disability
MeSH Terms: conditions — Stroke; Osteoarthritis, Knee; Agnosia

STUDY DESIGN:
Intervention Model Description: Two-arm parallel design where each group receives a distinct manual therapy intervention (SCS or MET) along with standardized physiotherapy. The study tracks changes in pain, ROM, and disability over 8 weeks.
Who Masked: Outcomes Assessor
Masking Description: Only the outcomes assessor was blinded to the participants' group assignments to ensure objective measurement of pain, ROM, and functional disability scores.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Strain Counterstrain with Routine Physical Therapy (Experimental): Participants in this arm received Strain Counterstrain (SCS) along with routine physical therapy. SCS involved identifying and holding tender points in positions of comfort for 90 seconds to relieve pain and improve range of motion. Routine physical therapy included TENS, infrared therapy, ultrasound, strengthening exercises (short arc quads, seated knee flexion/extension, terminal knee extension), and stretching exercises (straight leg raises, lying and sitting hamstring stretches). The intervention was delivered 5 days a week for 8 weeks. Education on weight management and joint protection strategies was also provided.
  Interventions: Behavioral: Strain Counterstrain with Routine Physical Therapy
- Muscle Energy Technique with Routine Physical Therapy (Experimental): Participants in this arm received Muscle Energy Technique (MET) along with routine physical therapy. MET involved post-isometric relaxation and slow eccentric isotonic stretching techniques targeting hamstrings and quadriceps, helping to restore joint mobility and muscle flexibility. Routine physical therapy included TENS, infrared therapy, ultrasound, strengthening exercises (short arc quads, seated knee flexion/extension, terminal knee extension), and stretching exercises (straight leg raises, lying and sitting hamstring stretches). The intervention was administered 5 days per week over 8 weeks, along with patient education on lifestyle and joint care.
  Interventions: Behavioral: Muscle Energy Technique with Routine Physical Therapy

INTERVENTIONS:
Behavioral: Strain Counterstrain with Routine Physical Therapy — This intervention involves applying the Strain Counterstrain (SCS) technique in combination with standard physical therapy. SCS targets tender points through passive positioning to reduce muscle tension and pain. The patient is positioned in a position of comfort for 90 seconds while monitoring the tender point. This is followed by gradual return to neutral. Routine physical therapy includes electrotherapy (TENS, IR, ultrasound), strengthening (short arc quads, terminal knee extension), and stretching exercises. The therapy is administered 5 days per week over 8 weeks.
  Arms: Strain Counterstrain with Routine Physical Therapy
Behavioral: Muscle Energy Technique with Routine Physical Therapy — This intervention combines Muscle Energy Technique (MET) with routine physical therapy. MET involves voluntary muscle contractions against resistance, followed by stretching to restore range of motion and relieve pain. Techniques include post-isometric relaxation and slow eccentric isotonic stretching, particularly targeting hamstring and quadriceps tightness. Routine physical therapy includes electrotherapy (TENS, IR, ultrasound), as well as structured strengthening and stretching exercises. The intervention was delivered 5 days a week for 8 weeks.
  Arms: Muscle Energy Technique with Routine Physical Therapy

SUMMARY:
This study aimed to evaluate the comparative effects of Strain Counterstrain (SCS) and Muscle Energy Technique (MET) on pain, range of motion (ROM), and functional disability in patients with knee osteoarthritis (KOA). Conducted as a single-blinded randomized control trial at the University of Lahore Teaching Hospital, 76 participants were divided into two groups, receiving either SCS or MET alongside routine physical therapy. Outcome measures included pain intensity, ROM, and functional disability via KOOS.

DETAILED DESCRIPTION:
This randomized controlled trial investigated the comparative efficacy of Strain Counterstrain (SCS) and Muscle Energy Technique (MET) in managing knee osteoarthritis (KOA) symptoms. A total of 76 patients meeting inclusion criteria were randomly assigned into two equal groups. Group A received SCS along with routine physical therapy, and Group B received MET with the same physiotherapy protocol. The interventions were carried out five days a week for eight weeks, and outcomes were measured at baseline, four weeks, and eight weeks. Pain was assessed using the Numeric Rating Scale (NRS), range of motion (ROM) via goniometry, and functional disability using the KOOS index.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 to 65 years (Pandiselvi, 2019).
* Patients who were willing and able to comply with the study protocol and follow-up procedures (Arslan et al., 2022).
* Patients having Grade 2 knee OA Kellgren and Lawrence system. In this system, grade 2 signifies minimal severity of OA (Ratzlaff et al., 2018).

Exclusion Criteria:

* Congenital deformities (Deng et al., 2021).
* Having any tumor or related pathology such as cancer (Arslan et al., 2022).
* Patients having any previous knee surgery (Khan et al., 2023).
* Patients with isolated/predominantly patellofemoral symptomatic osteoarthritis, inflammatory diseases, joint effusion, or excessive knee deformity (Deng et al., 2021).

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Pain intensity reduction measured by Numeric Pain Rating Scale (NPRS) | Baseline, Week 4, and Week 8
  Pain intensity was assessed using the Numeric Pain Rating Scale (NPRS), a validated 0-10 scale where 0 indicates "no pain" and 10 indicates "worst possible pain." Assessments were conducted at baseline, 4 weeks, and 8 weeks. A lower score represents improvement.

SECONDARY OUTCOMES:
Improvement in range of motion (ROM) measured using goniometry | Baseline, Week 4, and Week 8
  Range of motion (ROM) of the affected knee was measured using a standard universal goniometer. The focus was on knee flexion and extension. Measurements were taken at baseline, 4 weeks, and 8 weeks to evaluate changes over time.
Change in functional disability measured by KOOS questionnaire | Baseline, Week 4, and Week 8
  Functional disability was assessed using the Knee Injury and Osteoarthritis Outcome Score (KOOS). It includes five subscales (pain, symptoms, ADL, sport/recreation, QOL). Higher scores indicate better function. Assessed at baseline, 4 weeks, and 8 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Lahore Teaching Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ratzlaff C, Ashbeck EL, Guermazi A, Roemer FW, Duryea J, Kwoh CK. A quantitative metric for knee osteoarthritis: reference values of joint space loss. Osteoarthritis Cartilage. 2018 Sep;26(9):1215-1224. doi: 10.1016/j.joca.2018.05.014. Epub 2018 May 26. PMID 29842940